CLINICAL TRIAL: NCT05564910
Title: Computerized Cardiotocography and Fetal Heart Response to Maternal Coffee Intake: A Prospective Study
Brief Title: Computerized Cardiotocography and Maternal Coffee Habits
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco La Verde, Researcher, University of Campania Luigi Vanvitelli
Other Study IDs: 0018443/i
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Prenatal Care
Keywords: computerised cardiotocography; Fetal monitoring; nutrition in pregnancy; prenatal care; fetal heart rate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coffe group: Pregnant women who referred caffeine intake.
- Control group: Pregnant women without caffeine intake.

SUMMARY:
The study includes pregnant women referred for foetal antepartum computerized cardiotocography (cCTG) monitoring as outpatients. Pregnant women were divided into two groups based on their coffee intake: the coffee group and the control group. Each pregnant woman had cCTG. Two doctors assessed and recorded the amount of coffee taken by pregnant women before the CTG.

ELIGIBILITY:
Inclusion Criteria:

* gestationale age >37 weeks

Exclusion Criteria:

* fetal malformations,
* stillbirths
* preterm labour
* preterm and term premature rupture of membranes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: we included only term pregnant, who performed a computerized cardiotocography before the delivery.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Computerized cardiotocography | 1 day (cardiotocographic's test)
  Computerized cardiotocography (cCTG) parameters evaluate the fetal heart rate. We analyzed the cCTG between the two groups: pregnant who took coffee and pregnant with no coffee intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli studi della Campania "Luigi Vanvitelli"- OB & Gyn -, Napoli, Italia, Italy